CLINICAL TRIAL: NCT02340182
Title: The Role of the Microbiota in the Systemic Immune Response
Acronym: MISSION-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.J. Wiersinga, MD, PhD (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, W.J. Wiersinga, MD, PhD, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL42072.018.12; 2012_283 (Other: METC AMC)
Record Dates: First submitted 2013-07-08; First posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Healthy; Sepsis
Keywords: gut flora; antibiotics; systemic immune response; Volunteers
MeSH Terms: conditions — Sepsis | interventions — Vancomycin; Ciprofloxacin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antibiotics (Experimental): All volunteers will self-administer the following antibiotics for 7 consecutive days (concomitantly):
  1. Vancomycin 250mg 3dd2;
  2. Ciprofloxacin 500mg 2dd1;
  3. Metronidazole 500mg 3dd1.
  Interventions: Drug: Vancomycin; Drug: Ciprofloxacin; Drug: Metronidazole

INTERVENTIONS:
Drug: Vancomycin — 250mg 3dd2
Drug: Ciprofloxacin — 500mg 2dd1
Drug: Metronidazole — 500mg 3dd1

SUMMARY:
The objective of this study is to investigate the role of the gut microbiota in the systemic priming of immune effector cells. Twelve healthy male volunteers, 18-35 years of age, will be treated with broad spectrum antibiotics (ciprofloxacin, vancomycin, metronidazole) for seven days, in order to deplete the gut microbiota. Blood and faeces will be sampled before, 24 hours and 6 weeks after the 7-day period of antibiotics. Main study endpoints include laboratory parameters for inflammatory responses, functional assays (ex vivo stimulation assay) and gut microbiota composition.

DETAILED DESCRIPTION:
Rationale: Sepsis ranks among the top ten leading causes of death worldwide. Most nonsurvivors die in a state of immunosuppression. The gut microbiota exerts numerous beneficial functions in the host response against infections. Gut flora components express microorganism-associated molecular patterns (MAMPs) such as lipopolysaccharide (LPS), which are recognized by pattern recognition receptors (PRRs) expressed by neutrophils and macrophages. MAMPs from the intestinal microbiota constitutively translocate to the circulation and prime bone marrow derived neutrophils via PRRs. Antibiotic treatment, which is standard of care for all patients with sepsis, depletes the gut microbiota and leads to a diminished release of MAMPs and other bacteria derived products. This causes diminished priming of systemic immunity, which may attribute to sepsis associated immunosuppression and an increased susceptibility to invading bacteria.

Objective: To investigate the role of the gut microbiota in the systemic priming of immune effector cells

Study design: Within-subject-controlled intervention study in human volunteers

Study population: Twelve healthy male subjects, 18-35 years of age

Intervention: All subjects will be treated with broad spectrum antibiotics (ciprofloxacin, vancomycin, metronidazole) for seven days, in order to deplete the gut microbiota. Blood and faeces will be sampled before, 24 hours and 6 weeks after the 7-day period of antibiotics.

Main study parameters/endpoints: Laboratory parameters for inflammatory responses, functional assays (ex vivo stimulation assay) and gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male between 18 and 35 years of age
* Capable of giving written informed consent and able to comply with the requirements and restrictions
* Chemistry panel without any clinically relevant abnormality
* Normal defecation pattern (defined as <3x/ day and >3x/week)

Exclusion Criteria:

* Major illness in the past 3 months or significant chronic medical illness;
* History of any type of malignancy;
* Past or current gastrointestinal disease which may influence the gut microbiota;
* Known positive test for hepatitis C antibody, hepatitis B surface antigen or HIV;
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities;
* Use of tobacco products;
* History, within 3 years, of drug abuse;
* History of alcoholism and/or drinking more than 3 units of alcohol per day;
* The subject has received an investigational product within three months of day 1;
* Use of prescription or non-prescription drugs and herbal and dietary supplements within 6 months;
* Recent (< 12 months) use of antibiotics (any kind, except for dermal antibiotics);
* Allergy to antibiotics (any kind);
* Difficulty swallowing pills;
* Any other relevant issue.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Composite measure of Laboratory parameters for inflammatory responses. | up to 7 weeks
  Ex vivo response of whole blood, isolated monocytes or neutrophils to lipopolysaccharide.

OTHER OUTCOMES:
Side effects will be registered using a graded scale | up to week 7
A HITchip (human intestinal tract chip; 16S rRNA) analysis will be used to determine microbiome composition | up to week 7

CONTACTS AND LOCATIONS:
Overall Officials: Tom Van der Poll, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academisch Medisch Centrum, Amsterdam, North Holland, Netherlands